CLINICAL TRIAL: NCT02182297
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Doses (40 mg to 480 mg) of BI 201335 NA as Capsule(s) Administered to Healthy Male Subjects - a Randomised, Placebo-controlled (Within Dose Groups) and Double-blind Trial
Brief Title: Safety, Tolerability, and Pharmacokinetics of BI 201335 NA in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1220.13
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BI 201335 NA in single rising doses (Experimental)
  Interventions: Drug: BI 201335 NA in single rising doses
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 201335 NA in single rising doses
  Arms: BI 201335 NA in single rising doses
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this trial was to investigate safety, tolerability, and pharmacokinetics of BI 201335 ZW after administration of single rising doses from 40 mg to 480 mg of BI 201335 NA in healthy Japanese male volunteers.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be healthy male volunteers who meet the criteria below:

* Persons without clinically remarkable findings or clinically evident complications based on their concurrent illness, past medical history, physical examination, vital signs (blood pressure, pulse rate, and body temperature), 12-lead ECG, and laboratory test results
* Persons who are 20 or older and 35 or younger
* Persons with body mass index (BMI) of 18.5 kg/m2 or more and 25.0 kg/m2 less
* Persons who are willing to participate in this trial before study initiation and who give their written consent in accordance with the GCP (Good Clinical Practice)

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, body temperature, and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
* Prior history of jaundice
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of any drugs within 10 days prior to administration or during the trial
* Participation in another trial with an investigational product within four months prior to administration or during the trial
* Smoker (>10 cigarettes, >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days (during hospitalisation and end of trial)
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within 4 weeks prior to administration or during the trial)
* Excessive physical activities (within 1 week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of the trial site
* A history of additional risk factors for torsades de pointe (e.g., heart failure, hypokalemia, and family history of long QT syndrome)
* The use of concomitant medications that prolong the QT/corrected QT interval

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal findings in physical examination | Baseline and within 7 days after last trial procedure
Number of patients with clinically significant changes in vital signs (blood pressure, pulse rate) | Baseline, pre-dose and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose and day 12
Number of patients with abnormal findings in 12-lead electrocardiography (ECG) | Baseline, pre-dose and 1, 2, 4, 6, 8, 24, 48, 72 and 96 hours post-dose and day 12
Number of patients with abnormal changes in laboratory tests (haematology, clinical chemistry, and urinalysis) | Baseline, pre-dose and 24, 48, 72 and 96 hours post-dose and day 12
Number of patients with adverse events | up to day 12
Assessment of tolerability by the investigator on a 4-point scale | day 12 (within 7 days after last trial procedure)

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | pre-dose and 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
tmax (time from dosing to maximum concentration of the analyte in plasma) | pre-dose and 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
AUC0-∞ (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | pre-dose and 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | pre-dose and 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
λz (terminal elimination rate constant in plasma) | pre-dose and 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
t1/2 (terminal half-life of the analyte in plasma) | pre-dose and 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
MRTpo (mean residence time of the analyte in the body after po administration) | pre-dose and 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
CL/F (apparent clearance of the analyte in the plasma after oral administration) | pre-dose and 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Vz/F (apparent volume of distribution during the terminal phase λz following an oral administration) | pre-dose and 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) | 0-4, 4-12, 12-24, 24-48, 48-72 and 72-96 hours post-dose
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | 0-4, 4-12, 12-24, 24-48, 48-72 and 72-96 hours post-dose
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | 0-4, 4-12, 12-24, 24-48, 48-72 and 72-96 hours post-dose